CLINICAL TRIAL: NCT03417427
Title: A Multicenter Randomized Control Clinical Trail of Evaluating Effect of Demethylation Drug Combined With Chemotherapy in Patients With Intermediate-risk AML After Hematological Complete Remission
Brief Title: A Clinical Trail of Demethylation Drug Combined With Chemotherapy in Intermediate-risk AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuejie Jiang (Other)
Responsible Party: Sponsor-Investigator, Xuejie Jiang, Associate Professor, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LC2016YM005
Record Dates: First submitted 2017-05-13; First posted 2018-01-31 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Leukemia, Myeloid
Keywords: acute myeloid leukemia; Intermediate-risk; demethylation drug; complete remission
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Myeloid, Acute; Pathologic Complete Response | interventions — Decitabine; Cytarabine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decitabine and Ara-C (Active Comparator): Intermediate-risk AML patients with hematological complete remission and positive minimal residual disease (MRD) will receive decitabine (15mg/m2 d1-5) combined with high-dose of Ara-C (2g/m2 d4-6) consolidation chemotherapy.
  Interventions: Drug: Decitabine and Ara-C
- Ara-C (Placebo Comparator): Intermediate-risk AML patients with hematological complete remission and positive minimal residual disease (MRD) will receive high-dose of Ara-C (2g/m2 d4-6) consolidation chemotherapy.
  Interventions: Drug: Ara-C

INTERVENTIONS:
Drug: Decitabine and Ara-C — Decitabine in combination with high-dose of Ara-C is used to improve the effect of consolidation chemotherapy. It is expected to make minimal residual disease (MRD) become negative in more patients with intermediate-risk AML.
  Other Names: Decitabine in combination with high-dose of Ara-C
  Arms: Decitabine and Ara-C
Drug: Ara-C — Intermediate-risk AML patients with hematological complete remission and positive minimal residual disease (MRD) will receive high-dose of Ara-C (2g/m2 d4-6) consolidation chemotherapy.
  Other Names: High-dose of Ara-C
  Arms: Ara-C

SUMMARY:
It is often impossible to find therapeutic target in intermediate-risk AML, so it is very important to select appropriate chemotherapy protocol to eliminate minimal residual disease (MRD) in these AML patients. Recent studies demonstrated that leukemia microenvironment is the shelter nich for leukemia stem cells and the essential reason for impossibly eliminating MRD. Demethylation drug not only prove the effect of chemotherapy, but also change leukemia microenvironment through epigenetics modification. Both of them will result in eliminating MRD in patients with AML. The investigators designed a multicenter randomized control clinical trail to evaluate the effect of demethylation drug combined with chemotherapy in AML patients with intermediate-risk factors after hematological complete remission. Efficacy will be evaluated through MRD detected by flow cytometry every 1 month. Continuous negative MRD indicates a good prognosis. The patients with continuous negative MRD can select auto-HSCT or consolidation chemotherapy, those with continuous positive MRD should be considered as candidates of allo-HSCT. Overall survival and relapse free survival will be recorded after follow-up every 3 months. It will provide a basis for precision therapy and a new way for designing a novel protocol for intermediate-risk AML. This clinical trail will benefit to the AML patients with intermediate-risk factors.

ELIGIBILITY:
Inclusion Criteria:

* AML patients with normal heart, lung, liver and renal function, or without serious infection. ECOG score is below 2

Exclusion Criteria:

* AML patients with abnormal heart, lung, liver and renal function, or with serious infection. ECOG score is over 2

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease | 1 month
  Minimal residual disease is detected by flow cytometry every 1 month in AML patients.

SECONDARY OUTCOMES:
Overall survival | 3 months
  AML patients are followed up every 3 months to evaluate overall survival
Relapse free survival | 3 months
  AML patients are followed up every 3 months to evaluate relapse free survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital of Southern Medical University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided